CLINICAL TRIAL: NCT05619393
Title: Comparison of Kinematic Movements Between ACL Deficiency With ACL Reconstruction and Healthy People - Investigator Initiated Trial-
Brief Title: Comparison of Kinematic Movements Between ACL Deficiency With ACL Reconstruction and Healthy People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wang Joon Ho (Other)
Responsible Party: Sponsor-Investigator, Wang Joon Ho, MD, Professor, Department of Orthopaedic Surgery, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-05-019
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Reconstruction; Healthy People
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobilie Bi-planar X-ray Imaging system (Experimental)
  Interventions: Device: Mobilie Bi-planar X-ray Imaging system

INTERVENTIONS:
Device: Mobilie Bi-planar X-ray Imaging system — on the Mobilie Bi-planar X-ray Imaging system, images are acquired for three movements: walking, downhill walking, and squat

SUMMARY:
Comparison of kinematic movements between patients with anterior cruciate ligament rupture and post-operative patients and normal people using a mobile dynamic X-ray device.

DETAILED DESCRIPTION:
On a treadmill equipped with a mobile dynamic X-ray device, the subject will take three movements: walking, downhill walking, and squat, and the movement of the knee joint will be tracked. The investigators plan to quantify and compare the motion of the knee joint taken in patients with anterior cruciate ligament rupture, anterior cruciate ligament reconstruction, and normal people according to 6 degrees of freedom. Through this, the investigators plan to compare the functional instability between normal people and the ACL rupture patient group in daily life, and compare this with the ACL reconstruction patient group to see if surgery can reduce knee joint instability in everyday life. To confirm this, with mobile dynamic X-rays taken as the primary variable, the investigators took 1) normal subjects, 2) patients with anterior cruciate ligament rupture, 3) patients with more than 1 year after double bundle ACL reconstruction, and 4) single bundle anterior patients. the investigators plan to compare 6 degrees of freedom between patient groups who have had more than 1 year after cruciate ligament reconstruction and anterolateral ligament reconstruction. As secondary variables, the Lachman test and the Pivot shift test will be compared between the four groups.

ELIGIBILITY:
Inclusion Criteria

* Normal group

  1. Adults between 19 and 60 years of age
  2. Those who have no knee instability, locking, or jamming, and no history of surgery
  3. A person who has the will and ability to follow the procedures of this clinical trial protocol
  4. Those who voluntarily agreed in writing to participate in this clinical trial
* Anterior cruciate ligament rupture patient group

  1. Adults between 19 and 60 years of age
  2. Those with grade 3 or higher in the Lachmann test
  3. A person suspected of having an anterior cruciate ligament injury tear on magnetic resonance imaging (MRI)
  4. A person who has the will and ability to follow the procedures of this clinical trial protocol
  5. Those who voluntarily agreed in writing to participate in this clinical trial
* Patient group more than 1 year after anterior cruciate ligament reconstruction

  1. Adults between 19 and 60 years of age
  2. A person who has performed double bundle reconstruction; or Those who have performed single bundle reconstruction and anterolateral ligament reconstruction
  3. A person who has the will and ability to follow the procedures of this clinical trial protocol
  4. Those who voluntarily agreed in writing to participate in this clinical trial

Exclusion criteria

1. Those with degenerative arthritis of the knee joint
2. Those who need reoperation after anterior cruciate ligament rupture surgery, or those who have other knee surgery history, who are difficult to participate in the study under the judgment of the principal investigator
3. Patients with chronic inflammatory joint disease such as rheumatoid arthritis
4. Those whose growth plates are not closed
5. Patients who need companion surgery for ligament instability of grade II (grade 0: none, grade I: 0-5 mm, grade II: 5-10 mm, grade III: >10 mm) on physical examination
6. Pregnant and lactating women
7. Persons judged by other researchers as inappropriate for participation in clinical trials

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-07 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference for 6-Degree of freedom | Baseline
  Evaluate the difference in the result of measuring the six degrees of freedom of the knee joint, including the front and rear potentials of the knee joint, the inner and outer potentials, and the inner rotation/outer rotation.
  Measure the vertical distance between the femur posterior condyle and posterior tibia.
  The unit of measurement is millimeter .

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No